CLINICAL TRIAL: NCT04866004
Title: Feasibility and Impact of 28-days of Monitored Abstinence From Cannabis Use on Symptoms of Distress, Inflammation, and HIV Viral Load
Brief Title: Contingency Management for Cannabis Use for Persons With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Chukwuemeka Okafor, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-20-0886; K01DA047912 (NIH); HSC20220688H (Other: UT Health San Antonio)
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Marijuana; HIV Infections
MeSH Terms: conditions — Marijuana Abuse; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency Management - Cannabis (Experimental): Participants will be incentivized following biochemical verification (from urine samples) of cannabis abstinence.
  Interventions: Behavioral: Contingency Management - Cannabis

INTERVENTIONS:
Behavioral: Contingency Management - Cannabis — Participants in the contingency management program will be provided financial incentives for 28-days of cannabis abstinence. At every visit, participants will provide urine samples for the biochemical verification of cannabis abstinence). Participants with evidence of cannabis abstinence will be provided a financial incentive that increases across subsequent study visits.

SUMMARY:
The purpose of this study is to determine the feasibility and impact of 28-days of monitored abstinence from cannabis use on symptoms of depression and anxiety, pain, sleep, cannabis use withdrawal, HIV viral load and biomarkers of systemic inflammation among PLWH and who use cannabis regularly (weekly or more often). This will be a single arm pilot feasibility trial involving a contingency management program to induce cannabis abstinence. Specifically, the contingency management program will provide motivational (monetary) incentives to participants who achieve biochemically verified cannabis abstinence. Over the 28-days of this pilot feasibility trial, participants will attend seven study visits. During these visits, participants will complete survey questionnaires to assess sociodemographic, psychosocial, and behavioral factors. In addition, participants will provide blood and urine specimens for testing and quantitation of HIV viral load, biomarkers of systemic inflammation and for the detection of cannabis and other drugs of abuse.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive (confirmed via HIV medication or relevant HIV labs in subject's name)
* Self-report of cannabis use at least once per week in the 6-month period prior to consent
* Provide a positive urine toxicology (UTOX) screen for cannabis
* Not seeking treatment for cannabis use
* Willing to stop using cannabis for 28 days and attend eight study visits over six weeks.
* Ability and willingness to provide inform consent
* English fluency

Exclusion Criteria:

* Currently receiving treatment for cannabis or other drug use disorder
* Diagnosed or receiving treatment for a current major depressive or anxiety disorder
* Diagnosed with any current alcohol or substance use disorder (excluding nicotine) using the Structured Clinical Interview for Clinical Disorders (SCID) Interview (22)
* Positive UTOX screen for opioids
* Having a medical, psychiatric, occupational, or other condition that, in the judgment of the study physician, would make participation difficult or unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Sustained cannabis abstinence for 28-days | 28-days
  Cannabis abstinence will be defined as sustained reduction in quantitative levels of 11-Nor-9-carboxy-Δ⁹-tetrahydrocannabinol (THCCOOH) for 28-days

CONTACTS AND LOCATIONS:
Overall Officials: Chukwuemeka N Okafor, PhD, MPH, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Center for Neurobehavioral Research on Addiction, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT04866004/ICF_000.pdf